CLINICAL TRIAL: NCT06108778
Title: Adescriptive Study on Incidence of Metabolic Disorders in Neonatal Convulsions
Brief Title: Incidence of Metabolic Disorders in Neonatal Convulsions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Mohamed Sayed Ahmed, Assistant lecturer, Assiut University
Other Study IDs: Neonatal convulsions
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Neonatal Convulsions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — Investigations as CT,MRI.serum ammonia and lactate

SUMMARY:
Describe the incidence of metabolic disorders in neonatal convulsions affecting neonates at NICU Describe types of metabolic disorders causing neonatal convulsions

DETAILED DESCRIPTION:
Neonates are susceptible to seizures due to several physiologic factors and combination of risks that are uniquely associated with gestation, delivery,and the immediate postnatal period. Neonatal seizures can be challenging to identify therefore itis imperative that clinicians have ahigh degree of suspicion for seizures based on the clinical history or the presence of encephalopathy with or without paroxysmal abnormal movements. Acute symptomatic neonatal seizures are due to an acute brain injury, whereas neonatal onset_epilepsy may be due to underlying structural, metabolic ,or genetic disorders.Early identification and treatment are likely important for long term outcomes in acute symptomatic seizures though additional studies are needed to understand optimal seizure control metrics and the ideal duration of treatment. seizures may be the first and the major presenting feature of an inborn error of metabolism. seizures may be preceded by other major symptoms by areduced level of consciousness in achild with an organic acidemia or urea cycle defect or by loss of skills ,progressive weakness ,ataxia ,and upper motor signs in achild with lysosomal storage disorder or peroxisomal leukodystrophy.the metabolic causes of seizure vary according to age at presentation.

ELIGIBILITY:
Inclusion Criteria:

* Neonatal convulsions associated with vomiting,acidotic breathing,DCL,change of body tone or change in hair color
* Abnormal metabolic investigations (elevated serum ammonia and lactate ,persistent metabolic acidosis,abnormal metabolic screening and hypoglycemia
* persistent neonatal convulsions not respond to antiepileptic drugs

Exclusion Criteria:

* History of neonatal asphyxia
* History of birth trauma
* Signs of sepsis and CNS infection
* Neonate with electrolyte disturbance

Ages: 1 Day to 28 Days | Sex: All
Age Groups: Child
Study Population: Neonates with convulsions due to metabolic diseases
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2023-11-25 (Estimated); Primary Completion 2024-12-25 (Estimated); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
Describe incidence of metabolic disorders in neonatal convulsions affecting neonates at NICU | Baseline
  Describe types of metabolic disorders causing neonatal convulsions

REFERENCES:
- [Background] Russ JB, Simmons R, Glass HC. Neonatal Encephalopathy: Beyond Hypoxic-Ischemic Encephalopathy. Neoreviews. 2021 Mar;22(3):e148-e162. doi: 10.1542/neo.22-3-e148. PMID 33649088
- [Background] Stomnaroska O, Petkovska E, Jancevska S, Danilovski D. Neonatal Hypoglycemia: Risk Factors and Outcomes. Pril (Makedon Akad Nauk Umet Odd Med Nauki). 2017 Mar 1;38(1):97-101. doi: 10.1515/prilozi-2017-0013. PMID 28593892
- [Background] Balakrishnan U, Chandrasekaran A, Amboiram P, Ninan B, Ignatious S. Outcome of Inherited Metabolic Disorders Presenting in the Neonatal Period. Indian J Pediatr. 2021 May;88(5):455-462. doi: 10.1007/s12098-020-03522-6. Epub 2020 Oct 14. PMID 33051787